CLINICAL TRIAL: NCT00246480
Title: Pathogenesis of RSV Disease in the Elderly
Brief Title: RSV Disease in the Elderly
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0083
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2011-04

CONDITIONS: Respiratory Infections, Acute; Respiratory Syncytial Virus
Keywords: Respiratory Syncytial Virus Infections, RSV, elderly
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Respiratory syncytial virus (RSV) causes sickness and deaths in older people every winter. This study will investigate how aging affects the body's immune response (body's response to disease) to RSV. About 2000 people, age 21 and older, who reside in the upstate NY area, will be recruited. Two groups of subjects will be studied. The 1st group of volunteers will be recruited prior to the start of RSV season in year 1 of the study. These volunteers will include healthy people and people with various medical conditions. The 2nd group of volunteers will be patients admitted to Rochester General Hospital for acute respiratory illness. Procedures will include drawing blood from a vein in the arm (2 tablespoons), collecting nasal swabs, and collecting sputum. Volunteers may participate in study related procedures for up to 3 years.

DETAILED DESCRIPTION:
Respiratory infections account for significant excess morbidity and mortality among older people each winter. Influenza A virus and Respiratory Syncytial Virus (RSV) have emerged as two of the most important viruses for this age group. The resultant morbidity and mortality among these populations is substantial. Natural RSV infection in adults of various ages with mild, moderate, and severe RSV disease will be evaluated in order to accomplish the following primary objectives: to assess the effect of aging on the immune response to natural RSV infection; to assess the effect of aging on the clearance of RSV infection; to assess the effect of aging on the innate immune response to natural RSV infection; to assess the possibility of virus spread to the lower airways and; to assess the role of the RSV-specific immune response in the pathogenesis of severe disease. Study participants will include approximately 2000 persons, male and female, greater than or equal to age 21, including healthy persons, persons with common medical conditions (i.e., hypertension, diabetes, thyroid conditions, arthritis, coronary artery disease, skin cancer, etc), persons with underlying chronic pulmonary or cardiac conditions, and persons with signs and symptoms of acute respiratory tract illness who reside in the Upstate, New York area. A prospective cohort of ~800 persons will be recruited prior to the onset of RSV season in year one and followed for respiratory illnesses during each RSV season for three years or until the subject has a documented RSV illness. This group will contain persons of various ages and a spectrum of medical conditions. This population will be used to evaluate age-related differences in the immune response to RSV and viral shedding patterns.These volunteers are expected to provide primarily cases of mild to moderately severe RSV disease. A second group of subjects with signs and symptoms of acute respiratory tract illness will be recruited from the Lifetime After hours Urgent Care Center, Rochester General Hospital emergency room and inpatient medical service. Those identified with RSV infection will provide cases of moderate to severe RSV disease. At the end of RSV season, a control group will be selected. This group will be comprised from subjects chosen from the prospective cohort who did not have an RSV infection during that winter season. Controls will be matched by age and underlying conditions for each of the RSV infected subjects. The following outcome measures will be assessed: RSV severity: severe disease=hospitalized cases, mild-moderate disease=non-hospitalized cases; virus load: quantity and duration of RSV shedding as determined by quantitative RT-PCR; T cell responses; antibody: acute serum IgG to RSV F and G proteins by EIA and and neutralization titer to RSV A2 or B1 virus depending upon the infecting strain; local innate immune response: maximum IL-6 or IL-8 or MIP-1 alpha levels in nasal secretions; systemic innate immune response: maximum number of NK cells in the peripheral blood; and systemic inflammation: maximum serum IL-6 or C reactive protein value.

ELIGIBILITY:
Inclusion Criteria:

Prospective Cohort

* Greater than or equal to 21 years of age
* Able to provide written consent
* Telephone contact available
* Will reside in the Upstate New York area throughout the winter months

Hospital Cohort

* Greater than or equal to 21 years of age
* Able to provide written consent or legal guardian able to provide written consent
* Telephone contact available
* Symptoms of respiratory tract infection for less than or equal to 30 days duration. Symptoms can be all or any of the following: nasal congestion, cough, new or increased sputum or dyspnea, sore throat, with or without fever

Exclusion Criteria:

Prospective Cohort

* Known immunosuppressive condition including: HIV, active cancer currently receiving chemotherapy, hematological malignancy, autoimmune disorders.
* Documented RSV infection in the previous year
* Participation in previous RSV vaccine study

Hospital Cohort

* Known immunosuppressive condition including: HIV, active cancer currently receiving chemotherapy, hematological malignancy, autoimmune disorders.
* Symptoms of a respiratory infection for longer than 30 days.
* Participation in prior RSV vaccine study

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1401 (Actual)
Dates: Start 2005-10-03; Primary Completion 2008-05-28 (Actual); Study Completion 2008-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester General Hospital, Rochester, New York, United States